CLINICAL TRIAL: NCT00170989
Title: Comparison of the Combination of Valsartan 320 mg Plus Hydrochlorothiazide 12.5 mg and Valsartan 320 mg Plus Hydrochlorothiazide 25 mg to Valsartan 320 mg in Mild to Moderate Hypertensive Patients Not Adequately Controlled With Valsartan 320 mg
Brief Title: Valsartan/Hydrochlorothiazide Combination in Hypertensive Patients Not Controlled With Valsartan Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631C2302
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension
Keywords: hypertension; high blood pressure; valsartan; hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: valsartan plus hydrochlorothiazide

SUMMARY:
This study will test the effectiveness and safety of a combination treatment in patients whose blood pressure is not controlled with a single medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate hypertension

Exclusion Criteria:

* Severe hypertension
* History of stroke, myocardial infarction, heart failure, chest pain, abnormal heart rhythm
* Liver, kidney, or pancreas disease
* Insulin dependent diabetes
* Allergy to certain medications used to treat high blood pressure

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 2714 (Actual)
Dates: Start 2004-09; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure from baseline after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure from baseline after 8 weeks
Change from baseline in standing systolic and diastolic blood pressure after 8 weeks
Diastolic blood pressure less than 90 mmHg or at least a 10 mmHg decrease in diastolic pressure after 8 weeks
Diastolic blood pressure less than 90 mmHg after 8 weeks
Adverse events and serious adverse events at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland